CLINICAL TRIAL: NCT04894721
Title: Study of Efficacy and Safety of Ivermectin for COVID-19 Prophylaxis in Post-exposure Contact or Epidemiological Link
Brief Title: Prophylaxis for COVID-19: Ivermectin in Close Contacts of COVID-19 Cases (IVERNEX-TUC)
Acronym: IVERNEX-TUC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ministry of Public Health, Argentina (Other Government)
Responsible Party: Principal Investigator, Maria de los Angeles Peral de Bruno, Director of Research - Ministry of Health of Tucumán, Ministry of Public Health, Argentina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5077/410 CH 2020
Record Dates: First submitted 2021-05-06; First posted 2021-05-20 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: Ivermectin; Prophylaxis; COVID-19; Epidemiological link
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Randomized controlled. Experimental and Control Group in relationship of 2:1
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The EG receives ivermectin 0,6mg/kg of weight orally on days 1 (one) and 7 (seven) plus standard biosecurity care
  Interventions: Drug: Ivermectin
- Control Group (Placebo Comparator): The CG receives a placebo on days 1 (one) and 7 (seven) plus standard biosecurity care
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivermectin — 0,6mg/kg of weight orally on days 1 and 7
  Other Names: Iver
  Arms: Experimental Group
Other: Placebo — A substance with similar physical characteristics as ivermectin, without the active drug ingredient
  Arms: Control Group

SUMMARY:
Randomized controlled clinical trial on using oral ivermectin in COVID-19 prophylaxis supplying the drug to close contacts of confirmed cases.

DETAILED DESCRIPTION:
This is a randomized, double-blind, and controlled clinical trial that aims to evaluate the use of oral ivermectin in COVID-19 prophylaxis. The study has two arms in a relationship of 2:1: Experimental Group (EG n=500) and Placebo Group (CG n=250).

The sample size was calculated by applying a two-proportion comparison test. Type of two-sided test, 95% confidence or safety level (1-α), 95% statistical power, 75% P1 (proportion in the placebo group), 65% P2 (proportion in the new treatment or intervention group), size sample without adjustment (n = 543), 25% expected proportion of losses, n= 724 sample adjusted for losses.

The hypothesis of the study is that treatment with ivermectin may decrease the chance of occurrence/progress of clinical manifestations and onset of severe disease. Whereas control of the contagion on the first days of development of the disease, this treatment with ivermectin in suspected cases of COVID-19 (by epidemiological nexus) would contribute to the control of contagion at the first part of the infection, even in the absence of symptoms.

Categorical variables will be represented with frequencies and proportions, while continuous quantitative variables will be expressed as mean ± standard deviation (SD) or as median and interquartile range (IQR). The proportions will be compared using Pearson's Chi-square test or Fisher's exact test as appropriate, and continuous quantitative variables with Student's t test. The estimation of the efficacy of intensive treatment with Ivermectin will be calculated using Kaplan-Meier curves and the differences will be analyzed by means of the log-rank test. The risk will be calculated as a ratio of advantages for Intensive treatment with Ivermectin (Odds Ratio, OR) with its 95% confidence intervals (95% CI). A value of p <0.05 will be considered significant. Analyzes will be performed using Stata 11.2 software.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years either sex
* Women of childbearing age with a negative pregnancy test
* In close contact group or epidemiological nexus of a positive COVID-19 case
* Able to understand and grant informed consent
* Real-time - polymerase chain reaction test with a negative result

Exclusion Criteria:

* Known hypersensitivity or allergy to any component of the drug under evaluation
* Age under 18 years
* Use of immunosuppressants (including systemic corticosteroids) in the last 30 days
* Pregnant or lactating
* Patients with other acute infectious diseases
* Patients with autoimmune disease and/or chronic decompensated diseases
* Who have received a vaccine for COVID-19 (1/2 dose) or that have taken ivermectin (prior to 30 days of the study) or who are participating in another COVID-19 prophylaxis study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects who were diagnosed with COVID-19 in EG and CG (Negative polymerase chain reaction - real-time). | At 2 weeks
  Pearson's Chi-square and proportion test

SECONDARY OUTCOMES:
Contagion risk. | Up to 2 weeks
  Odd Ratio
Prophylactic effect associated with patient's preexisting comorbidity | Up to 2 weeks
  Logistic regression test

CONTACTS AND LOCATIONS:
Overall Officials: Rossana Chahla, Ph. D, Principal Investigator — Ministry of Public Health, Tucumán, Argentina
Locations (1):
- SI.PRO.SA, Ministerio de Salud Pública, San Miguel de Tucumán, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chong CR, Sullivan DJ Jr. New uses for old drugs. Nature. 2007 Aug 9;448(7154):645-6. doi: 10.1038/448645a. No abstract available. PMID 17687303
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Ahmed S, Karim MM, Ross AG, Hossain MS, Clemens JD, Sumiya MK, Phru CS, Rahman M, Zaman K, Somani J, Yasmin R, Hasnat MA, Kabir A, Aziz AB, Khan WA. A five-day course of ivermectin for the treatment of COVID-19 may reduce the duration of illness. Int J Infect Dis. 2021 Feb;103:214-216. doi: 10.1016/j.ijid.2020.11.191. Epub 2020 Dec 2. PMID 33278625
- [Background] Ahmed Elgazzar, Basma Hany, Shaimaa Abo Youssef et al. Efficacy and Safety of Ivermectin for Treatment and prophylaxis of COVID-19 Pandemic, 13 November 2020, PREPRINT (Version 1) available at Research Square [https://doi.org/10.21203/rs.3.rs-100956/v1]
- [Background] Hirsch RR, Carvallo, Héctor E. Ivermectin as Prophylaxis Against COVID-19 Retrospective Cases Evaluation. Microbiol Infect Dis. 2020; 4(4): 1-8.

DOCUMENTS (2):
  • Study Protocol (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT04894721/Prot_002.pdf
  • Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT04894721/ICF_003.pdf